CLINICAL TRIAL: NCT03202901
Title: Accute Effect of B-Turmactive Both on Mild and Moderate Knee Pain on Healthy Volunteers: a Pilot, Randomised, Parallel and Double Blind Pilot Trial
Brief Title: Accute Effect of B-Turmactive Both on Mild and Moderate Knee Pain on Healthy Volunteers
Acronym: TURMACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: Hospital Universitari Sant Joan de Reus (Other); University Rovira i Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-TURMACTIVE
Record Dates: First submitted 2016-12-12; First posted 2017-06-29 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Knee Injuries; Inflammation Knees
Keywords: knee-pain, curcuma, inflammation
MeSH Terms: conditions — Knee Injuries; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B-turmactive (Experimental): 1 pill of B-turmactive: 500 mg hydrosoluble fraction (free curcuminoid fraction) + 19.5 mg of lipid soluble fracion (curcuminoids enriched) + 22.5 mg vitamin C.
  Interventions: Dietary Supplement: B-turmactive
- Placebo (Placebo Comparator): Yeast brew extract (200 mg)
  Excipients:
  120 mg cellulose (food additive E-460) 40 mg Compritol® E ATO (food additive E-471) 4 mg Magnesium stearate (food additive E-572)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: B-turmactive — The treatment consists of daily administration of B-TURMACTIVE®.
  Treatment with B-TURMACTIVE® will last 7 days to determine the effects of the product in the short term, during which the volunteers will be visited 4 times:
  V0 screening: to evaluate the inclusion and exclusion criteria. V1 inclusion and randomisation (Day 1): 1st day treatment and intervention. Measure primary and secondary variables V2 (Day 3): the primary endpoint will be monitored by telephone (perception of pain).
  V3 (Day 7): Day 7 of treatment and final intervention. Measure primary and secondary variable
  Arms: B-turmactive
Dietary Supplement: Placebo — The treatment consists of daily administration of placebo capsule with identical format and harmless thant B-turmactive product.
  Treatment with placebo will last 7 days to determine the effects of the product in the short term, during which the volunteers will be visited 4 times:
  V0 screening: to evaluate the inclusion and exclusion criteria. V1 inclusion and randomisation (Day 1): 1st day treatment and intervention. Measure primary and secondary variables V2 (Day 3): the primary endpoint will be monitored by telephone (perception of pain).
  V3 (Day 7): Day 7 of treatment and final intervention. Measure primary and secondary variable
  Arms: Placebo

SUMMARY:
The goal of this study is to assess the short (acutte) effect of B-Turmactive (one week treatment) both on mild/moderate knee pain

DETAILED DESCRIPTION:
Join pain is a common cause of consultation in primary health care in the adult population. Indeed, people who suffer knee pain, mostly due to osteoarthritis, require analgesic treatment, often with some secondary effects. Therefore, the research to find a natural and efficient product to reduce knee pain in a short period of time, facilitating recovery after exercise and without side effects have an interest both for industry and for the general population.

B-turmactive is an extract of Curcuma longa mixing two fractions in a single product: a) soluble fraction free-curcuminoids but rich in polysaccharides and b) curcuminoids fraction with cyclodextrin. Both fractions plus vitamin C are B-turmactive.

Previous preclinical studies suggest that B-turmactive could exert an acute effect in healthy people that suffer mild or moderate knee pain and, furthermore could reduce inflammation process.

Therefore, the goal of this study is to assess the short (acute) effect of B-Turmactive (one week treatment) both on mild/moderate knee pain

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 30 and 65 years old.
* Score between 15-25 out of 50 within WOMAC pain subscale
* Signed informed consent.

Exclusion Criteria:

* people who take concomitant drug or supplements (multivitamins) that could interfere with the product under study.
* people who suffer froma arthritis of the knee.
* people who take more than two analgesic drugs and/or anti-inflammatory for more than three months.
* people who have a history of surgery or trauma affecting the knee.
* people with gluten sensitivity and/or allergy to gluten and sulphites (the placebo containing yeast).
* people with anemia (haemoglobin ≤ 13g/dL in men and ≤ 12g/dL in women).
* people with BMI ≥ 30 kg / m
* women pregnant or breastfeeding.
* women with menopausal suffering from osteoporosis.
* people with liver abnormalities (ALT, AST), kidney (creatinine) or other muscular issues (creatine kinase).
* people with neurological disorders.
* people who have participated in a clinical trial or intervention study the last 30 days prior to inclusion in the study.
* people unable to follow the guidelines of the study.
* people who not signed the informed consent.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC pain subscale | 1 week (day 1; day 3; day 7)
  Visual analogue scale of 5 items derived from 24 items WOMAC scale

SECONDARY OUTCOMES:
Anthropometric data | 1 week (day 1;day 7)
  Trained dieticians measure weight and body composition using a body composition analyzer (Tanita SC 330-S; Tanita Corp., Barcelona, Spain) and height using a well mounted stadiometer (Tanita Leicester Portable; Tanita Corp., Barcelona, Spain), to calculate BMI: weight/height x height (kg/m2).
  Waist circumference (cm) is measured midway between the lowest rib and the iliac crest using an anthropometric tape.
Biochemistry for on-going study control | 1 week (day 1;day 7)
  Aspartate aminotransferase (AST) (IU/L), Alanine aminotransferase (ALT) (IU/L), Tryglycerides (mg/dL), total Cholesterol (mg/dL), High-density lipoprotein cholesterol (HDL-c) (mg/dL), Low-density lipoprotein cholesterol (LDL-c) (mg/dL) and Glucose (mg/dL).
  Total cholesterol, HDL-c, Tryglicerides, AST, ALT and glucose are measured in serum by standardized enzymatic automated methods in a PENTRA-400 autoanalyzer (ABX-Horiba Diagnostics, Montpellier, France). LDL-c is calculated by the Friedewald formula.
Inflammatory markers | 1 week (day 1;day 7)
  C reactive protein (mg/dL), IL-1β (ng/mL), IL-6 (ng/mL), Prostaglandin E metabolite (PGEM) (ng/mL) are measured in serum and determined by standardized methods in a Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain) or using a specific ELISA kit.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Valls, PhD, Study Director — University Rovira i Virgili; Rosa Solà, MD, PhD, Principal Investigator — Hospital Universitari Sant Joan, Universitat Rovira i Virgili, CTNS; Anna Pedret, PhD, Study Chair — University Rovira i Virgili; Elisabet Llauradó, PhD, Study Chair — University Rovira i Virgili; Montse Giralt, MD, PhD, Study Chair — University Rovira i Virgili
Locations (1):
- Technological Center of Nutrition and Health (CTNS), Reus, Spain